CLINICAL TRIAL: NCT04030039
Title: Cohort Study of Clinical Outcomes in Chronic HBV Infection Patients With Low HBsAg Loads Under Unplanned Intervention
Brief Title: Cohort Study of Clinical Outcomes in Chronic HBV Infection Patients With Low HBsAg Under Unplanned Intervention
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Head of liver diseases center, Beijing Ditan Hospital
Other Study IDs: DTXY017
Record Dates: First submitted 2019-06-22; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Chronic Hepatitis B Infection
Keywords: Chronic hepatitis B; interferon; nucleotide; HBV; HBsAg; HBV DNA
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Interferons

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- chronic hepatitis B patients during the immune control period: Patients with chronic HBV infection during the immune control period do not have any clinical treatment intervention cohort
- Therapy group A: After chronic hepatitis B patients were treated with interferon, HBsAg level of these patients < 100 IU / ml, and they continued to be treated with interferon
  Interventions: Drug: Interferon
- Therapy group B: After chronic hepatitis B patients were treated with interferon, HBsAg level of these patients < 100 IU / ml, and they stopped to be treated with interferon
  Interventions: Drug: Interferon
- Therapy group C: After chronic hepatitis B patients were treated with interferon, HBsAg level of these patients < 100 IU / ml, and they continued to be treated with sequential nucleoside analogues
  Interventions: Drug: Interferon; Drug: nucleoside analogues
- Therapy group D: After chronic hepatitis B patients were treated with nucleoside analogues, HBsAg level of these patients < 100 IU / ml, and they continued to be treated with sequential interferon
  Interventions: Drug: Interferon; Drug: nucleoside analogues
- Therapy group E: After chronic hepatitis B patients were treated with nucleoside analogues, HBsAg level of these patients < 100 IU / ml, and they continued to be treated with the nucleoside analogues
  Interventions: Drug: nucleoside analogues

INTERVENTIONS:
Drug: Interferon — chronic hepatitis B patients with interferon therapy
  Groups: Therapy group A; Therapy group B; Therapy group C; Therapy group D
Drug: nucleoside analogues — chronic hepatitis B patients with interferon therapy
  Groups: Therapy group C; Therapy group D; Therapy group E

SUMMARY:
All chronic hepatitis B (CHB) patients were diagnosed and treated in the liver disease department of the Hepatology Center of Beijing Ditan Hospital affiliated to Capital Medical University and those who received antiviral therapy (interferon and nucleoside analogues) reached HBsAg<100 IU/ml. The enrolled subjects were divided into the following six observation cohorts: 1) CHB patients in the immunological control period, without any clinical treatment intervention; 2) After interferon therapy, HBsAg<100 IU/ml, continued interferon therapy; 3) After interferon therapy, HBsAg<100 IU/ml, stopped interferon treatment; 4) After interferon therapy, HBsAg<100 IU/ml, sequential nucleoside analog treatment; 5) After nucleoside analogue treatment, HBsAg<100 IU/ml, sequential interferon treatment; 6) After treated with nucleoside analogues, HBsAg<100 IU/ml, continuing the nucleoside analog treatment. The follow-up observation period was 96 weeks under non-planned intervention. During the observation period, HBV indicators and biochemical indicators, serum AFP and liver imaging (liver ultrasound) were examined regularly. The main evaluation index was the incidence of HBsAg disappearance during the observation period. Secondary evaluation indicators: the rate of HBV DNA turning positive, the rate of HBeAg turning positive and hepatitis incidence. To observe the inactive carrier status of low HBsAg content and the incidence of HBsAg disappearance, clinical outcomes and influencing factors in patients with CHB under different antiviral interventions.

DETAILED DESCRIPTION:
This study is a clinical observational cohort study. All chronic hepatitis B patients were diagnosed and treated in the liver disease department of the Hepatology Center of Beijing Ditan Hospital affiliated to Capital Medical University and those who received antiviral therapy (interferon and nucleoside analogues) reached HBsAg<100 IU/ml. The enrolled subjects were divided into the following six observation cohorts: 1) chronic Hepatitis B patients in the immunological control period, without any clinical treatment intervention in this cohort; 2) After interferon therapy, HBsAg<100 IU/ml, continued interferon therapy in this cohort; 3) After interferon therapy, HBsAg<100 IU/ml, stopped interferon treatment in this cohort; 4) After interferon therapy, HBsAg<100 IU/ml, sequential nucleoside analog treatment in this cohort; 5) After nucleoside analogue treatment, HBsAg<100 IU/ml, sequential interferon treatment in this cohort; 6) After treated with nucleoside analogues, HBsAg<100 IU/ml, continuing the nucleoside analog treatment in this cohort. The follow-up observation period was 96 weeks under non-planned intervention. During the observation period, HBV DNA loads, HBsAg/anti-HBs, HBeAg/anti-HBe and biochemical indicators, serum AFP and liver imaging (liver ultrasound) were examined regularly. The main evaluation index was the incidence of HBsAg disappearance during the observation period. Secondary evaluation indicators: the rate of HBV DNA turning positive, the rate of HBeAg turning positive and hepatitis incidence. To observe the inactive carrier status of low HBsAg content and the incidence of HBsAg disappearance, clinical outcomes and influencing factors in patients with CHB under different antiviral interventions.

ELIGIBILITY:
Inclusion Criteria:

* Inactive carrier status and chronic hepatitis B (CHB) patients with anti-viral therapy (interferon and nucleoside analogues) reaching HBsAg < 100 IU/ml.

Exclusion Criteria:

* coinfection with other viruses including HCV, HDV, and HIV;
* syphilis antibody positive;
* co-exist other liver diseases including alcoholic liver disease, metabolic liver disease, fatty liver, drug induce liver injury, and autoimmune liver disease;
* complication of cirrhosis or liver cancer.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis B patients with HBsAg < 100 IU/ml in an inactive carrying state were enrolled and treated with antiviral therapy (interferon and nucleoside analogs). All patients with chronic hepatitis B infection were eligible for the diagnostic criteria of the Chinese Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2015).
Sampling Method: Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of HBsAg disappearance during the 96-week study in different observation cohorts | 96 weeks
  The incidence of HBsAg disappearance during the 96-week study in different observation cohorts

SECONDARY OUTCOMES:
HBV DNA re-yang rate during the 96-week study period in different observation cohorts | 96 weeks
  HBV DNA re-yang rate and HBeAg re-yang rate during the 96-week study period in different observation cohorts
HBeAg re-yang rate during the 96-week study | 96 weeks
  HBeAg re-yang rate during the 96-week study

OTHER OUTCOMES:
liver cancer during the 96-week study period in different observation cohorts Incidence | 96 weeks
  liver cancer during the 96-week study period in different observation cohorts Incidence
Hepatitis episodes during the 96-week study period in different observation cohorts Incidence | 96 weeks
  Hepatitis episodes during the 96-week study period in different observation cohorts Incidence
cirrhosis decompensation during the 96-week study period in different observation cohorts Incidence | 96 weeks
  cirrhosis decompensation during the 96-week study period in different observation cohorts Incidence
its complications during the 96-week study period in different observation cohorts Incidence | 96 weeks
  its complications during the 96-week study period in different observation cohorts Incidence

CONTACTS AND LOCATIONS:
Overall Officials: Yao Xie, Principal Investigator — Beijing Ditan Hospital, Beijing, China
Locations (1):
- liver disease center, Beijing Ditan Hospital, Beijing, Beijing Municipality, China